CLINICAL TRIAL: NCT05482321
Title: Contrast Enhanced Ultrasound Imaging of Pancreas Blood Flow in type1 Diabetes
Brief Title: Pancreas Ultrasound Imaging in type1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1543
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type1diabetes; Insulitis; Pancreas Inflamed
Keywords: ultrasound; tissue perfusion; contrast; diabetes; pancreas
MeSH Terms: conditions — Pancreatitis; Diabetes Mellitus | interventions — Injections; perflutren

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: SOP (healthy) subjects. Part I of study (optimizing protocol).
  Interventions: Drug: Definity Suspension for Injection
- Group 2: Control (healthy and autoantibody positive) subjects. Part II of study (cross-sectional study)
  Interventions: Drug: Definity Suspension for Injection
- Group 3: T1D subjects. Part II of study (cross-sectional study)
  Interventions: Drug: Definity Suspension for Injection

INTERVENTIONS:
Drug: Definity Suspension for Injection — * DEFINITY is administered as per manufactures instructions
  * 1 vial of DEFINITY is allowed to warm to room temperature and activated by 45s shaking on a VIALMIX
  * Withdraw the activated milky white suspension using the provided Dispensing Pin, PINSYNC or 18-20 gauge syringe needle, from the middle of the liquid in the inverted vial.
  * Deliver a dose of 10 μl/kg of 'milky white suspension' IV as a bolus, delivered over 30seconds.
  * Following imaging, provide a 10 mL flush of preservative-free saline
  * Wait at least 30minutes until second dose (if provided).
  Other Names: DEFINITY

SUMMARY:
The overall goal of this study is to develop and test a novel method involving ultrasound imaging, in order to detect the development of type 1 diabetes. In this study the investigators will first establish a standard operating procedure for measuring pancreas blood flow speed and volume in the pancreas of human subjects. The investigators will then determine 1) whether these pancreas blood flow factors differ between healthy subjects and those who have recently developed type1 diabetes; and 2) how variable measurements are in healthy subjects and subjects that recently developed type1 diabetes, both between subjects and over time. To address these aims the investigators will perform pancreas ultrasound measurements in each subject using an approved injectable 'bubble' contrast agent that allows measurement of pancreas blood flow. The investigators will compare ultrasound measurement with characteristics of the subject's type 1 diabetes, including genetic factors, glucose levels and other circulating factors, as well as other factors that may influence blood flow in the pancreas independent of type1 diabetes. The successful conclusion of this study will indicate whether measuring pancreas blood flow speed/volume will be helpful in monitoring whether type1 diabetes will emerge and thus will allow a large scale study to answer this question.

DETAILED DESCRIPTION:
Study Design and Research Methods

Part I:

5 subjects from SOP group Goal: Optimize settings for destruction-replenishment contrast-enhanced ultrasound scan

1. Subject recruited at the Barbara Davis Center
2. Subject provides written consent
3. Review medical history (exclusion if required)
4. Subject refrains from eating for ~6h prior to measurement
5. Subject visits University of Colorado Hospital CTRC echo lab
6. CTRC staff places peripheral intravenous line (PIV)
7. Research staff collects vital signs, height and weight
8. Subject received conventional ultrasound scan to locate pancreas tail (by Sonographer, verified by radiologist).
9. Subject receives DEFINITY dose
10. Subject receives destruction-replenishment contrast-enhanced ultrasound scan (adjust settings to optimize)
11. Pause for 30 minutes, allowing subject to stand and move
12. Repeat steps 9-11 (once).
13. Subject de-identified.
14. Analyze data.

Part II:

30 subjects from control group (healthy controls and multiple islet autoantibody positive subjects), 15 subjects from T1D group.

Goal: characterize subject variability and test whether healthy subjects and those with T1D show differing contrast measures

1. Subject recruited at the Barbara Davis Center
2. Subject provides written consent
3. Review medical history (exclusion if required)
4. Subject refrains from eating for ~6h prior to study
5. Subject visits University of Colorado Hospital CTRC echo lab
6. Subject completes questionnaire (family history of diabetes, exclusion criteria)
7. CTRC staff places peripheral intravenous line (PIV)
8. Research staff collects vital signs, height and weight
9. Subject received conventional ultrasound scan to locate pancreas tail (by Sonographer, verified by radiologist).
10. Subject receives DEFINITY dose
11. Subject receives destruction-replenishment contrast-enhanced ultrasound scan (under SOP)
12. Pause for 30 minutes, allowing subject to stand and move
13. Repeat steps 10-12 (once).
14. Subject de-identified
15. Analyze data.

In part I a single repeat measurement may be made to aide in the optimization of data collection. In part II a single repeat measurement is made to assess short-term intra-subject measurement variability.

In part I and part II, a subject will be asked to return on a separate date (within 1 year of the initial scan) for a repeat procedure using an additional DEFINITY delivery method (bolus or infusion, whichever was not given at the initial visit) or if data collection was not of sufficient quality during the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female age 18-65
* Ability and willingness of patient to participate fully in all aspects of this clinical study
* Written informed consent obtained and documented

Exclusion Criteria:

* Excessive body size preventing effective scan of the pancreas as determined by sonographer
* Evidence of exocrine pancreatic disease, including pancreatitis, cystic fibrosis, pancreatic adenocarcinoma, or neuroendocrine tumor.
* Subjects who are pregnant or breast-feeding
* Subjects incapable of giving assent/informed written consent
* Known or suspected hypersensitivity to perflutren
* Known history or suspected unstable cardiopulmonary conditions (acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure, or serious ventricular arrhythmias)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 subjects will be healthy subjects who will receive contrast-enhanced ultrasound 'destruction-replenishment' measurements, in order to optimize and establish the standard operating procedure (SOP) for this measurement in the pancreas of human subjects. This SOP will then be applied to Group 2 (healthy subjects and autoantibody positive subjects) and Group 3 (recent onset type1 diabetes) subjects as part of the cross-sectional study. Classification of type 1 diabetes includes meeting ADA criteria for diabetes, within 180 days of diagnosis, and evidence of at least 1 islet-associated autoantibody.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Primary outcome 1 | End of part I (6 months)
  Optimized a contrast-enhanced ultrasound 'destruction-replenishment' protocol for imaging pancreas blood flow kinetics in adult human subjects.
Primary outcome 2 | End of part II (1 year)
  Comparison of pancreas blood flow kinetics (i.e. 'destruction-replenishment' k2 'reperfusion rate' parameter) between control and T1D subjects.
Primary outcome 3 | End of part II (1 year)
  Determining inter-subject variability in pancreas blood flow kinetics (i.e. the 'destruction-replenishment' k2 'reperfusion rate' parameter) among control subjects and among T1D subjects
Primary outcome 4 | End of part II (1 year)
  Determining reproducibility in the measurement of pancreas blood flow kinetics (i.e. the 'destruction-replenishment' k2 'reperfusion rate' parameter) within subjects. This will initially focus on short-term intra-subject measurement variability.

SECONDARY OUTCOMES:
Secondary outcome 1 | End of part II (1 year)
  Comparison between control and T1D subjects for other parameters resulting from the measurement of pancreas blood flow kinetics (i.e. the 'destruction-replenishment' 'reperfusion amplitude' A, 'destruction efficiency' 1-B and 'pre-destruction signal' parameters).
Secondary outcome 2 | End of part II (1 year)
  Determining inter-subject variability among control subjects and among T1D subjects for other parameters resulting from the measurement of pancreas blood flow kinetics (i.e. the 'destruction-replenishment' 'reperfusion amplitude' A, 'destruction efficiency' 1-B and 'pre-destruction signal' parameters).
Secondary outcome 3 | End of part II (1 year)
  Correlation of pancreas blood flow kinetics with blood glucose and HbA1c (to test for a link between the measurement and glucose control).
Secondary outcome 4 | End of part II (1 year)
  Comparison of pancreas blood flow kinetics with HLA haplotype or whether subject has first-degree relative with T1D (to test for a link between the measurement and T1D genetic risk).
Secondary outcome 5 | End of part II (1 year)
  Comparison of pancreas blood flow kinetics with subject BMI, age, heart rate, blood pressure (to test for a link between the measurement and subject characteristics)
Secondary outcome 6 | End of part II (1 year)
  Assessment of subject autoantibodies, c-peptide levels (to ensure subjects free of diabetes do not have islet autoimmunity and to ensure subjects with T1D have islet autoimmunity and residual beta cell mass)

CONTACTS AND LOCATIONS:
Overall Officials: Richard KP Benninger, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No